CLINICAL TRIAL: NCT01538342
Title: Role of Tyrosine Kinase Lyn and Cleaved Form by Caspases in Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-API-03
Record Dates: First submitted 2012-01-13; First posted 2012-02-24 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Psoriasis; Atopic Dermatitis
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- chronic plaque psoriasis (Other): 3 biopsies: 2 lesional and 1 non-lesional
  Interventions: Other: 3 Biopsies
- pustular psoriasis (Other): 3 biopsies: 2 lesional and 1 non-lesional
  Interventions: Other: 3 Biopsies
- erythrodermic psoriasis (Other): 3 biopsies: 2 lesional and 1 non-lesional
  Interventions: Other: 3 Biopsies
- atopic dermatitis (Other): 2 biopsies: 1 lesional and 1 non-lesional
  Interventions: Other: 2 biopsies
- healthy patients (Other): 1 biopsy of healthy skin.
  Interventions: Other: biopsy

INTERVENTIONS:
Other: 3 Biopsies — 3 biopsies: 2 lesional and 1 non-lesional
  Arms: chronic plaque psoriasis; erythrodermic psoriasis; pustular psoriasis
Other: 2 biopsies
  Other Names: 1 lesional and 1 non-lesional
  Arms: atopic dermatitis
Other: biopsy — 1 biopsy ok healthy skin
  Arms: healthy patients

SUMMARY:
Psoriasis is a chronic autoimmune disorder of the skin. In this disease, the inflammatory caspases, cysteine proteases involved in the processing of many proteins, are activated. Transgenic mice expressing the cleaved form of caspases by Lyn, a tyrosine kinase Src family, develop an inflammatory syndrome with the characteristics of human psoriasis.

To clarify the relationship between the cleaved form of Lyn by caspases and psoriasis, the investigators intend to develop a clinical study to analyze the expression, cleavage and activity of Lyn and the activation of caspases from skin biopsies of patients with this disease.

This study will be conducted on a cohort of patients with different forms of psoriasis (plaque, pustular and erythrodermic) and atopic dermatitis, another skin disorder associated with chronic inflammation. Thus, the investigators will evaluate the expression and activity of Lyn from skin lesion (L) and non-lesional (NL) from the same patient in parallel with the level of caspase activation and apoptotic inflammatory.

Thus, the investigators will verify that the cleavage by caspases of Lyn is associated specifically with psoriasis, as the investigators believe, or more generally to the skin inflammation. The investigators work would then define the cleavage by caspases of Lyn as a new potential marker of human psoriasis.

ELIGIBILITY:
Inclusion Criteria:

Psoriasis arms:

* Plaque psoriasis and erythrodermic more than 10% of body surface area.
* Pustular psoriasis of at least 1% of body surface.

  * Atopic dermatitis arm:Patients with atopic dermatitis has been identified and inflammatory lesions on the skin.
  * Healthy arm:People not suffering from any skin disease

Exclusion Criteria:

* Systemic treatment of psoriasis for at least 4 weeks and / or local treatment for at least 2 weeks at the time of study entry.
* Patient with significant infection and / or immunocompromised.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Cleavage of Lyn | 1 day
  The cleavage of Lyn will be determined in the different extracts of skin of patients with western blotting using an antibody specific for Lyn recognizing the native form but also the form cleaved by caspases.
Expression levels of Lyn | 1 day
  The expression levels of Lyn and its cleaved form will be quantified using the software MultiGauge. The investigators will also determine the level of activity of Lyn using an antibody directed against the active form phosphorylated. The level of expression of proteins of interest will be reported at the level of protein expression control (ERK2) whose expression does not vary depending on the samples (load control).
Specific activity of apoptotic caspases 3, 6, 7, 8 and 9, and inflammatory caspases 1, 4, and 5 | 1 day
  The investigators will determine the specific activity of apoptotic caspases 3, 6, 7, 8 and 9, and inflammatory caspases 1, 4, and 5 test microplate. The principle of this test is based on the use of a specific substrate of caspases coupled to a fluorochrome that fluoresces when it is released after the action of caspase-level target aspartate. The fluorescence emission, which is proportional to the amount of active caspase in the sample is then measured with a fluorometer.

SECONDARY OUTCOMES:
Development of a monoclonal antibodyspecific for the cleaved form of caspases by Lyn | 1 day
  Development of a monoclonal antibody specific for the form cleaved by caspases of Lyn. Once obtained and validated, this tool will be especially useful for immunohistological analysis of Lyn on skin sections from patients with psoriasis. Then we can also analyze which skin cells express preferentially cleaved form of Lyn.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul ORTONNE, PU-PH, Study Director — Centre Hospitalier Universitaire de Nice; Sandrine MARCHETTI, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France; Marie-Aleth RICHARD, PU-PH, Principal Investigator — AP-HM; Carle PAUL, PU-PH, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - Assistance Publique - Hôpitaux de Marseille, Marseille
  - University Hospital of Nice, Nice
  - University Hospital of Toulouse, Toulouse

REFERENCES:
- [Derived] Aira LE, Goncalves D, Bossowski JP, Rubio-Patino C, Chiche J, Paul-Bellon R, Mondragon L, Gesson M, Lecucq-Ottavi P, Obba S, Colosetti P, Luciano F, Bailly-Maitre B, Boyer L, Jacquel A, Robert G, Ricci JE, Ortonne JP, Passeron T, Lacour JP, Auberger P, Marchetti S. Caspase 1/11 Deficiency or Pharmacological Inhibition Mitigates Psoriasis-Like Phenotype in Mice. J Invest Dermatol. 2019 Jun;139(6):1306-1317. doi: 10.1016/j.jid.2018.11.031. Epub 2018 Dec 17. PMID 30571969
- See also: Related Info — http://www.unice.fr/c3m/FR/Equipe1.html